CLINICAL TRIAL: NCT03860727
Title: Role of iExaminer as Teaching Aid for Direct Ophthalmoscopy
Brief Title: Comparison of Ophthalmoscopy Findings Using PanOptic vs PanOptic + iExaminer
Status: Completed | Type: Observational
Sponsor: State University of New York at Buffalo (Other)
Collaborators: Welch Allyn (Industry)
Responsible Party: Principal Investigator, Andrew L Reynold, Clinical Assistant Professor, State University of New York at Buffalo
Other Study IDs: STUDY00002262
Record Dates: First submitted 2018-09-13; First posted 2019-03-04 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Vision Disorders
MeSH Terms: conditions — Vision Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Diagnostic Test: Welch Allyn IExaminer — Fundus Examination

SUMMARY:
To examine how helpful the iExaminer will be as a training aid for medical students. The investigators will look into whether 1) it helps the medical students find pertinent eye findings for certain diagnoses and 2) it improves the medical students comfort level compared to using the PanOptic alone.

DETAILED DESCRIPTION:
Direct ophthalmoscopy is a vital skill for screening emergent conditions as well as chronic ocular pathologies for nonophthalmic physicians. Many eye care practitioners are first exposed to this tool during their medical education and are expected to have a certain degree of proficiency with it down the line. This skill requires practice, however, and given that there is a limited amount of time and exposure, it is not surprising that there is a general lack of familiarity and confidence among students and physicians with using the direct ophthalmoscope (Gilmour et al.,2017; Schulz et al., 2014; Day et al.,2017).

A myriad of techniques and models have attempted to change this and improve the efficacy in teaching direct ophthalmoscopy. Studies have shown that students prefer learning how to use the direct ophthalmoscope with human subjects rather than simulators, and that the students prefer using fundus photographs to learn important diagnostic findings over the ophthalmoscope (Kelly et al.,2013). There have also been studies comparing the direct ophthalmoscope to the PanOptic, which gives a fixed working distance from the patient and a larger field of view (Day et al.,2017). These studies have noted more "ease of use" and accuracy in using the PanOptic among first year medical students and physicians (McComiskie et al.,2004; Petrushkin et al., 2012). New technological advances such as the iExaminer application have also been recently introduced, allowing the eye care physicians to take fundus images on their smart phone using a smart phone application and attachment to the PanOptic. Studies have shown the iExaminer application is able to produce "clinically adequate" fundus images (Day et al.,2017).

From the literature review, there have not been any studies that compare the PanOptic alone versus the PanOptic with the iExaminer application as an introductory teaching tool for medical students. The iExaminer will not only allow the user to utilize the view obtained from the PanOptic, but also allow an instructor to observe and help coach the user on relevant findings and take pictures for future reference or instruction. This provides a potentially effective learning device which can help users accurately identify more relevant ophthalmic findings. The investigators also believe that this will help increase the medical students confidence level and encourage them to practice with these devices again at future opportunities.

ELIGIBILITY:
Inclusion Criteria:

- All second-year medical students at the University at Buffalo Jacobs School of Medicine and Biomedical Sciences may be included in our final study sample.

Exclusion Criteria:

* Students who have had significant prior exposure to direct ophthalmoscopy (e.g. they have used the direct ophthalmoscopy, PanOptic, or PanOptic with the iExaminer on a regular basis for more than one week).
* Students with poor enough visual acuity that will prevent them from doing direct ophthalmoscopy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Second-year medical students at the University at Buffalo Jacobs School of Medicine and Biomedical Sciences attending Ophthalmoscopy class as a part of required didactic sessions. Volunteering patients with normal or eye pathology will be recruited for students to perform Ophthalmoscopy with PanOptic and iExaminer
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-08-28 (Actual); Primary Completion 2019-05-07 (Actual); Study Completion 2019-05-07 (Actual)

PRIMARY OUTCOMES:
Students confidence in using iExaminer to diagnose fundus findings | 9 months
  Students will be provided with survey questions to assess their confidence level in accurately diagnosing fundus findings using iExaminer combined with Panoptic vs Panoptic alone

SECONDARY OUTCOMES:
Students comfort in using iExaminer combined with Panoptic vs Panoptic alone | 9 months
  The fundus findings diagnosed by students using panoptic with be compared to when students used iExaminer attached to Panoptic

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Reynolds, MD, Principal Investigator — The Ira G. Ross Eye Institute - University at Buffalo; Pimpiroon Ploysangam, Principal Investigator — The Ira G. Ross Eye Institute - University at Buffalo
Locations (1):
- The Ira G. Ross Eye Institute, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No